CLINICAL TRIAL: NCT03166969
Title: Predictors of Occult Atrial Fibrillation in 171 Patients With Cryptogenic TIA and Minor Stroke
Acronym: HOLTER-21J
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Pr Fernando PICO, Investigator coordinator, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P14/08_HOLTER 21J
Record Dates: First submitted 2016-09-12; First posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Cryptogenic Transient Ischemic Attack and Minor Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients taken care in neurovascular unit (Experimental)
  Interventions: Procedure: Holter 21 days

INTERVENTIONS:
Procedure: Holter 21 days

SUMMARY:
Retrospective study, single-center, on 171 patients, presented a cryptogenic TIA and Minor stroke.

This study objective is to determine profitability of Holter 21 days for screening paroxystic ACFA / flutter in cryptogenic TIA/Minor stroke, and identify the predictive factors of discovery a paroxystic ACFA on Holter 21 days. Clinical and échocardiographics factors, and brain imaging (scanner and MRI) will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Cryptogenic TIA/Minor stroke
* Age > 18 years
* Medical care in Neuro Vascular Unit of CH Versailles
* Holter 21 days performed

Exclusion Criteria:

1. ACFA history
2. ECG or telemetry who showed ACFA before the Holter initializing
3. Carotid Stenosis / symptomatic vertebral
4. Arterial dissection
5. Prothrombotic state demonstrated by laboratory tests
6. Infective endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2007-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number of atrial fibrillation detected on long duration ( 21 days) cardiac rythm holter monitoring | Day 21
  Atrial fibrillation >= 30 secondes

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Versailles, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sudacevschi V, Bertrand C, Chadenat ML, Tarnaud C, Pico F. Predictors of Occult Atrial Fibrillation in One Hundred Seventy-One Patients with Cryptogenic Transient Ischemic Attack and Minor Stroke. J Stroke Cerebrovasc Dis. 2016 Nov;25(11):2673-2677. doi: 10.1016/j.jstrokecerebrovasdis.2016.07.014. Epub 2016 Aug 2. PMID 27495831